CLINICAL TRIAL: NCT05651269
Title: Milciclib in Combination With Gemcitabine in Advanced Non-Small Cell Lung Cancer
Brief Title: Milciclib in Combination With Gemcitabine in Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILS-020
Record Dates: First submitted 2022-12-02; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Milciclib plus gemcitabine (Experimental): Name: milciclib Dose: 150 mg/day Mode of administration: oral
  Combination product:
  Name: gemcitabine Dose: 1000 mg/m2 Mode of administration: intravenous
  Interventions: Drug: Milciclib Dose: 150 mg/day Mode of administration: oral

INTERVENTIONS:
Drug: Milciclib Dose: 150 mg/day Mode of administration: oral — milciclib plus gemcitabine
  Other Names: Combination product: gemcitabine Dose: 1000 mg/m2 Mode of administration: intravenous

SUMMARY:
The goal of this interventional clinical study is to evaluate the safety and efficacy of Milciclib plus gemcitabine in the treatment of persons with advanced NSCLC. This is an open label uncontrolled clinical trial

Eligible patients will receive 150 mg/day of milciclib orally using the 7 days on/7 days off schedule in combination with gemcitabine at the dose of 1000 mg/m² on Days 1, 8, and 15 every 4 weeks. Treatment cycles will be repeated every 4 weeks until progressive disease (radiologic or symptomatic deterioration), the start of a new systemic anticancer therapy, unacceptable toxicity, withdrawal per investigator's judgment, or withdrawal of consent, whichever occurs first.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, non-randomized, open-label, single-arm Phase 2 study in locally advanced non-resectable recurrent and/or metastatic KRAS-mutated NSCLC after failure of at least 1 line of SoC therapy.

All patients will be screened for KRAS mutation status. A total of up to 28 patients harboring G12A, G12D, G12F, G12R, G12S, G12V, or G13D KRAS mutations, or, any pathogenic KRAS mutation other than G12C mutations will be enrolled and treated. According to the Simon's 2-stage design, 13 patients will be treated at Stage 1 with up to 15 patients treated at Stage 2.

At the completion of Stage 1, a review of the tumor response evaluation will be undertaken to determine if the second stage should be conducted. If there are 2 or more patients with a complete response (CR) or partial response (PR) in the first 13 patients, an additional 15 patients will be accrued.

Stage 1 will be considered complete when all patients have experienced progressive disease (radiologic or symptomatic deterioration), started a new systemic anticancer therapy, have withdrawn per investigator's judgment or experienced unacceptable toxicity, have withdrawn consent, or have completed 6 cycles of treatment.

In addition, Stage 1 patients who, at the time of transition to Stage 2, were responding with a CR, PR, or stable disease, will be allowed to continue in the study at the recommended Phase 2 dose; or lower for safety reasons). These patients will not be part of the 15 new patients to be targeted in Stage 2, because they will have already received treatment with milciclib plus gemcitabine in Stage 1, but they will provide additional safety information regarding prolonged treatment with milciclib plus gemcitabine

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC with an associated G12A, G12D, G12F, G12R, G12S, G12V, or G13D KRAS mutation, or, any pathogenic KRAS mutation other than G12C, as determined by a Sponsor-approved laboratory
* Male or female patients at least 18 years of age
* Advanced unresectable recurrent or metastatic disease not amenable to local treatment with surgery or radiotherapy
* Documented disease progression after at least one line of prior SoC therapy
* Presence of measurable disease on computed tomography (CT) or magnetic resonance imaging (MRI) scan as defined by RECIST v1.1. A previously irradiated lesion may be considered a target lesion if clearly progressing
* Previous systemic anticancer treatment completed ≥ 3 weeks, major surgery ≥ 2 weeks, and radiation therapy ≥ 4 weeks prior to study enrollment
* Any adverse effects from prior surgery, radiotherapy, or antineoplastic therapy must have improved to Grade 1 or less by the time of enrollment
* ECOG performance status 0-2 at the time of enrollment
* Life expectancy at least 12 weeks
* Adequate bone marrow function as evidenced by meeting all the following requirements:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/μL without the use of hematopoietic growth factors within the last 2 weeks before screening
  * Platelet count 100,000 cells/μL without the use of platelet transfusion within the last 2 weeks before screening
  * Hemoglobin ≥ 9 g/dL without the use of red blood cell (RBC) transfusion within the last 2 weeks before screening
* Adequate hepatic function as evidenced by meeting all the following requirements:

  * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), unless explicitly related to documented Gilbert's syndrome
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3 × ULN; if liver metastases are present, then ≤ 5 × ULN is allowed
  * Adequate renal function as evidenced by an estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2 of body surface area.
* Female patients of childbearing potential (FCBP) must present with a negative serum pregnancy test and must agree to employ adequate birth control measures for the duration of the study and until 3 months after the end of last dose of the study drug. Female patients who are lactating must agree to stop breastfeeding from the start of study treatment until 1 month after the end of treatment. Lack of childbearing potential is indicated by > 12 months without menses, or after surgical sterility, or as indicated by follicle-stimulating hormone (FSH) concentration.
* Male patients must be surgically sterile or agree to use a double-barrier contraception method or abstain from heterosexual activity with an FCBP starting at the first dose of treatment and until 3 months after the last dose of the study drug. Male patients must also agree to refrain from sperm donation, storage, or banking during these same time periods.
* Patient is willing and able to comply with the requirements of the study protocol.

Exclusion Criteria:

* Previous treatment with sotorasib or any experimental anti-KRAS targeted agent, and/or previous treatment with gemcitabine
* Documented KRAS G12C mutation and previously untreated with sotorasib
* Existing Grade 2 or higher retinal conditions (e.g., retinal tear, exudate, hemorrhage)
* Existing Grade 2 or higher neurological condition (tremor, ataxia, hypotension, confusion)
* Significant intercurrent illnesses and/or any of the following:

  * Active uncontrolled peptic ulcer disease
  * Uncontrolled seizure disorders
  * Active and uncontrolled CNS metastases (indicated by clinical symptoms, cerebral edema, corticosteroid and/or anticonvulsant requirement, or progressive disease); for controlled CNS metastases, patient should have been off corticosteroids for at least 14 days or on a tapering or stable dose of corticosteroids at a maximum dose of 12 mg/day prednisone-equivalent, without overt evidence of significant neurological deficits prior to enrollment
* Significant cardiac conduction abnormalities, including known familial prolonged QT syndrome, or screening QTcF > 480 msec
* Symptoms of congestive heart failure Grade 2 or higher
* Active, uncontrolled bacterial, fungal, or viral infection or an unexplained fever > 38.5°C which in the investigator's opinion might compromise the patient's participation in the study
* Known history of difficulty swallowing, malabsorption, or other conditions that may reduce absorption of the product
* Chronic Grade ≥ 2 diarrhea
* Presence or history of any other active malignancy within 2 years other than a history of adequately treated basal or squamous cell carcinoma of the skin, or any adequately treated in situ carcinoma
* Active known human immunodeficiency virus ( HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Active hepatitis B is defined as positive hepatitis B surface antigen (HBsAg) or immunoglobulin (Ig)M hepatitis B core antibody (anti-HBc) with or without positive HBV DNA. Active hepatitis C is defined as positive HCV RNA and/or anti-HCV antibody. HIV test according to local practice and local regulatory guidance
* Female patient who is pregnant or lactating at the time of enrollment
* Any other medical or social condition deemed by the investigator to be likely to interfere with a patient's ability to cooperate and participate in the study or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Disease progression | The study will be closed 6 months after the last scheduled visit
  The primary endpoint is an independent, central reader-assessed, blinded to time of scan, and confirmed objective response rate (ORR), defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR), using RECIST v1.1. Any patient with CR or PR must be able to confirm the CR or PR at least 4 weeks following the first observation.

SECONDARY OUTCOMES:
Duration of response | time from date of randomization to date of death from any cause or end of study up to 12 months
  The secondary efficacy endpoints (using central reader-assessed response according to RECIST v1.1 when applicable) are:
  * Duration of response (DoR), defined as the duration between first documentation of CR or PR to first documentation of disease progression or death
  * Progression-free-survival (PFS), defined as the time from the date of first dose of study drug to the date of first documented disease progression or death due to any cause
  * Time to response (TTR), defined as the time from first dose of study drug to first documentation of CR or PR
  * Overall survival (OS), defined as the time from the date of first dose of study drug to the date of death due to any cause
Adverse Events | Up to 6 months after the last scheduled visit
  Incidence of AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Study Chair — Tiziana Life Sciences

IPD SHARING:
Plan to Share IPD: No
There is no planned sharing of data